CLINICAL TRIAL: NCT00724724
Title: The Effectiveness and Safety of Butylphthalide Soft Capsules in Secondary Prevention of Ischemic Stroke Trial
Acronym: ESCAPE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Liying Cui, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2006BAI01A10-3
Record Dates: First submitted 2008-07-26; First posted 2008-07-29 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Stroke; Transient Ischemic Attack
Keywords: Stroke; Transient Ischemic Attack
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Butylphthalide Soft Capsules + Aspirin
  Interventions: Drug: Butylphthalide Soft Capsules
- 2 (Active Comparator): Aspirin
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Butylphthalide Soft Capsules — Butylphthalide Soft Capsules: 2 tablets Bid for 1 year Aspirin: 100mg for 1 year
  Other Names: Butylphthalide Soft Capsules, En Bi Pu (NBP)
  Arms: 1
Drug: Aspirin — Aspirin 100mg Qd for 1 year
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of Butylphthalide Soft Capsules (En Bi Pu, NBP) in Secondary Prevention of Ischemic Stroke

DETAILED DESCRIPTION:
The efficacy and safety of Butylphthalide Soft Capsules (En Bi Pu, NBP)in acute ischemic stroke has been demonstrated in China recently. Its role in secondary prevention of ischemic stroke need to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic cerebral infarction or TIA within 90 days.
2. Aged above 40 years old.
3. Cranial CT or MRI scan exclude intracranial hemorrhagic diseases
4. Stable clinical and neurological conditions.
5. Informed consent is obtained.

Exclusion Criteria:

1. Intracranial hemorrhage
2. Stroke of other unkonwn causes, or other known causes, such as Takayasu arteritis, Moyamoya disease, dissecting aneurysm and hypercoagulable state, carotid endarterectomy, angiogram, or cardiac surgery
3. Cardio embolism
4. Patients with anticoagulants treament including heparin or warfarin
5. Severe co-morbid or unstable medical condition, ie, heart failure, respiratory failure and renal failure, severe liver dysfunction, malignancy with likelihood of death within the next 2 years
6. Significant memory or behavioural disorder, ie, Alzheimer disease, etc, daily care needed.
7. A Modified Rankin score is more than 4
8. Abnormal liver function: ALT or AST level >1.5 times upper limit of normal; Abnormal renal function: serum creatinine level >2.0mg/dl or 177umol/l:
9. Concurrent participation in another clinical trial
10. Uncontrolled hypertension : systolic blood pressure greater than 180mmHg, or diastolic blood pressure greater than 100mmHg
11. Haemostatic disorder or thrombocytopenia (i.e., PLT<100×109/l).
12. Currently active peptic ulcer disease
13. Pregnant or breast feeding
14. Planned for major surgery, carotid endarterectomy, or carotid angioplasty
15. Unable to give informed consent.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2008-08; Primary Completion 2011-06 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Newly onset ischemic stroke | 1 year follow up
vascular events including newly onset TIA,intracerebral hemorrhage,myocardic infarction,unstable angina pectoris, occlusion of peripheral artery | 1 year follow up
Small vessel disease defined by white matter lesions on MRI | 1 year follow up

SECONDARY OUTCOMES:
All-cause death | 1 year follow up

CONTACTS AND LOCATIONS:
Locations (49):
- China (49):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hosptial, Beijing, Beijing Municipality
  - China Pla General Hospital, Beijing, Beijing Municipality
  - Beijing Daxing District Hospital, Beijing, Beijing Municipality
  - Beijing Ji Shui Tan Hospital,the 4Th Medical College of Peking University, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - China Rehabilition Research Center, Beijing, Beijing Municipality
  - General Hospital of Navy, Beijing, Beijing Municipality
  - Luhe Hospital of Tongzhou Distict Beijing, Beijing, Beijing Municipality
  - No 263 Hospital of Pla, Beijing, Beijing Municipality
  - No 309 Hospital of Pla, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Pinggu County Hospital Beijing, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Daping Hospital, Chongqing, Chongqing Municipality
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - Guangzhou First Municipal People'S Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital,Sun Yat-Sen Unversity, Guangzhou, Guangdong
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Yutian County Hospital, Yutian, Hebei
  - Hebei North University, Zhangjiakou, Hebei
  - The First Hospital of Harbin Medical University, Harbin, Helongjiang
  - The Second Hospital of Harbin Medical University, Harbin, Helongjiang
  - Henan Provincial People'S Hospital, Zhengzhou, Henan
  - The Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Xiangya Hospital of Centre-South University, Changsha, Hunan
  - Inner Mongolia Baotou City Central Hospital, Baotou, Inner Mongolia
  - The Appurtenant Hospital of Chifeng University, Chifeng, Inner Mongolia
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing General Hospital of Nanjing Military Command, Nanjing, Jiangsu
  - The Affiliated Drumtower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jilin University, Changchun, Jilin
  - The Third People'S Hospital of Dalian, Dalian, Liaoning
  - The First Affiliated Hospital of China Medical Sciences University, Shenyang, Liaoning
  - Qinghai Provincial People'S Hospital, Xining, Qinghai
  - Qilu Hospital of Shangdong University, Jinan, Shandong
  - The Second Hospitalof Shangdong University, Jinan, Shandong
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - West China Center of Medical Sciences, Chengdu, Sichuan
  - The General Hospital Under Tianjin Medical Sciences University, Tianjin, Tianjin Municipality
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Xinjiang Medical University, Uramuqi, Xinjiang Uygur Autonomous Region
  - Second Affiliated Hospital Zhejiang University College of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang